CLINICAL TRIAL: NCT04442217
Title: Factors Associated With Adherence to Hygiene-related Behaviors and Viral Mitigation Protocols During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Omid V. Ebrahimi, Mr., University of Oslo
Other Study IDs: REK125510-11
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Adherence to WHO-advised Hygiene-related Behavior; Adherence to Viral Mitigation Protocols
MeSH Terms: interventions — Prospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Prospective study with two measurement points investigating the impact of viral mitigation protocols on mental health — Prospective study with two measurement points investigating the impact of viral mitigation protocols on mental health

SUMMARY:
Study description:

The preset study seeks to investigate factors associated with of hygiene-related behaviors and adherence to viral mitigation protocols during the COVID-19 pandemic. In particular, factors associated with of adherence to WHO-advised hygiene-related behaviors and adherence to governmental mitigation protocols are investigations.

The aim of the project is to:

* Inform the policymakers, the general public, scientists, and health practitioners about the cognitive, behavioral, emotional, motivational, and trait components underlying hygiene-related behaviors and adherence.
* Help policymakers better understand adherence and the factors it is associated with, providing empirical grounds to advance societies battle against the COVID-19-virus from an epidemiological perspective by promoting factors that increase adherence.

Hypothesis/Research questions Hypothesis 1: Risk perception, altruism and governmental trust will significantly be associated with both adherence and hygiene-related behavior, with increased risk perception, altruism, and governmental trust associated with higher rates of adherence and hygiene-related behavior. The personality traits conscientiousness and agreeableness will significantly be associated with both adherence and hygiene related behavior, with increased conscientiousness, and agreeableness associated with higher rates of adherence and hygiene-related behavior. Furthermore, beliefs about pandemic protocol efficacy and beliefs about collective mitigation behavior (i.e., "it is only useful to follow transmission protocols if everyone else does") will be associated with adherence to viral mitigation protocols and hygiene-related behaviors.

Research Question 1: Is there a difference between the use of various platforms to obtain information about COVID with regards to adherence to viral mitigation protocols and hygiene-related behaviors? Research Question 2: To what extend are different sources of obtaining information associated with adherence to hygiene-related behavior and adherence to viral mitigation protocols? Research Question 3: To what extent are different personality traits (measured with the Short Big Five Inventory-10 (BFI-10)) associated with adherence to viral mitigation protocols and hygiene-related behaviors?

DETAILED DESCRIPTION:
Hypothesis/Research questions Hypothesis 1: Risk perception, altruism and governmental trust will significantly be associated with both adherence and hygiene-related behavior, with increased risk perception, altruism, and governmental trust associated with higher rates of adherence and hygiene-related behavior. The personality traits conscientiousness and agreeableness will significantly be associated with both adherence and hygiene related behavior, with increased conscientiousness, and agreeableness associated with higher rates of adherence and hygiene-related behavior. Furthermore, beliefs about pandemic protocol efficacy and beliefs about collective mitigation behavior (i.e., "it is only useful to follow transmission protocols if everyone else does") will be associated with adherence to viral mitigation protocols and hygiene-related behaviors.

Research Question 1: Is there a difference between the use of various platforms to obtain information about COVID with regards to adherence to viral mitigation protocols and hygiene-related behaviors? Research Question 2: To what extend are different sources of obtaining information associated with adherence to hygiene-related behavior and adherence to viral mitigation protocols? Research Question 3: To what extent are different personality traits (measured with the Short Big Five Inventory-10 (BFI-10)) associated with adherence to viral mitigation protocols and hygiene-related behaviors?

Statistical analyses:

Two hierarchical regression analyses will be conducted: one with adherence to hygiene-related behavior as the dependent variable, and the second with adherence to pandemic protocols as the dependent variable. In both hierarchical regression analysis, the first step will include the demographic characteristics (control variables) age, gender, and education. The second step will include risk perception, altruism, governmental trust, personality traits (i.e., neuroticism, extroversion-introversion, openness, conscientiousness, agreeableness), beliefs about pandemic protocol efficacy and beliefs about collective mitigation behavior.

Part correlations will be reported, presenting the effect size of the hypothesized predictors on adherence, revealing the most important variables related to adherence behavior. Multicollinearity and other statistical assumptions will be checked using examined. Multicollinearity will be assessed with common guidelines (VIF < 5 and Tolerance > 0.2; Hocking, 2003; O'Brian, 2007).

All analyses and questions addressed in the forthcoming paper that are not pre-specified in this pre-registered protocol will be defined as exploratory.

Sensitivity analyses and random subsample replications of the main findings will be conducted following selection of a random sample of participants that ensure a proportionate ratio between the collected sample and the adult population of Norway.

Possible transformations:

All variables will be assessed in their original and validated format as is recommended practice, as long as this is possible with regards to statistical assumptions underlying the pre-defined analyses (i.e., multiple regression). However, if this is not possible with regards to the statistical assumptions behind the analyses, transformation (e.g., square root or log-transformations) may be needed to apply interval-based methods. The investigators will examine the degree of skewness and evaluate this against the assumptions and analyses before choosing the appropriate analysis. The pre-registered and planned analyses include multiple regression as long as the assumptions underlying these analyses are met. Alternatively, a non-parametric test will be used.

Inference criteria Given the large sample size in this study, the investigators pre-define their significance level: p < 0.01 to determine significance.

Sample size and power calculation:

The present study is part of a larger project with the first part aiming to investigate predictors of adherence through regression analyses, and the second part aiming to examine directional relations amongst specific symptoms and their centrality through complex systems approaches (i.e., network analysis). Consequently, power calculations are based on power required for network analyses. Following power analysis guidelines by Fried & Cramer (2017), it is recommended that the number of participants are three times larger than the number of estimated parameters. However, more conservative recommendations by Roscoe (1975) for multivariate research, recommends sample size that is ten times larger than the number of estimated parameters. Thus, following these two approaches respectively, between 1395 to 4650 participants are required. Data will be collected for three weeks, and participants are based on a representative and random sample of Norwegian adults, randomly selected and provided equal opportunity to partake in the study, providing digital consent.

Missing data:

The TSD system (Services for Sensitive Data), a platform used in Norway to store person-sensitive data verifies participants officially through a kind of national ID number to give them full right to withdraw their data at any time, following the European GDPR (General Data Protection Regulation) laws. Accordingly, participants are allowed to withdraw their own data at any time. The survey includes mandatory fields of response. Participation is voluntarily, and withdrawal of provided data is possible at any moment. The investigators do not expect participants to withdraw their data and thus expect no missing data. However, if participants do withdraw their data, The investigators will conduct state-of-art missing data analyses and investigate whether data is missing at random.

Variables:

Outcome measures: as described in primary outcome measures section: 1) adherence to viral mitigation protocols; and 2) adherence to WHO-recommended hygiene-related behaviors.

Predictors: All 5 Big Five Personality Traits are measured by the validated Brief Version of the Big Five Personality Inventory (BFI-10). Risk perception is measured with a three-item measure adapted for the COVID-19 pandemic, querying about the perceived risk of the COVID-19 virus for 1) oneself; 2) other individuals; and 3) society at large. Governmental trust is measured with a single item adapted for the COVID-19 pandemic, querying about the whether one trusts in the governments judgements and decisions concerning handling of the pandemic. Altruism is measured with a single item adapted for the pandemic, querying about personal importance given to helping society and peers. Beliefs about protocol efficacy and beliefs about collective mitigation behavior are both measured with single items adapted for the COVID-19 pandemic, querying about beliefs concerning the efficacy of initiated protocols against the pandemic and beliefs about perceived usefulness of adhering when a proportion of others do not.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical NPIs, and
* Who provide digital consent to partake in the study.

Exclusion Criteria:

* Children and adolescents (individuals below 18)
* Adults not residing in Norway during the measurement period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Biological Sex and self-representation of gender are measured
Study Population: All adults above 18 years residing in Norway and thus experiencing identical mitigation protocols are invited to participate the study, reaching randomly online with an equal opportunity of participating.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
Adherence to WHO-advised hygiene-related | Data is set to be collected starting from 22nd of June until enough data has been collected. The data collection period will last no longer than three weeks.
  Adherence to WHO-advised hygiene related behavior is measured with 7 items querying about hygiene-related behavior as recommended by the WHO, measured with on a 5-point likert scale, measuring the frequency of these behaviors for the past month (0 = not at all to 4 = Every day)
Adherence to viral mitigation protocols | Data is set to be collected starting from 22nd of June until enough data has been collected. The data collection period will last no longer than three weeks.
  o Adherence to viral mitigation protocols is measured with 5 items querying about adherence to mitigation protocols initiated by the Norwegian government, measured with on a 5-point likert scale, measuring the frequency of adherence to these protocols for the past month (0 = not at all to 4 = Every day).

CONTACTS AND LOCATIONS:
Overall Officials: Omid V. Ebrahimi, Double PhD Candidate, Principal Investigator — University of Oslo; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo; Asle Hoffart, PhD, Principal Investigator — Modum Bad